CLINICAL TRIAL: NCT04726644
Title: Ventral Hernias in Cirrhotic Patients
Brief Title: Evaluation of Surgical Techniques in Cirrhotic Patients With Ventral Hernias
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Abu Elfatth, Al-rahji University Hospital, Faculty of Medicine, Assiut, Egypt, Assiut University
Other Study IDs: El-rajhi Liver Hospital
Record Dates: First submitted 2021-01-23; First posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Ventral Hernias in Cirrhotic Patients
MeSH Terms: interventions — Herniorrhaphy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients: cirrhotic patients with ventral hernia
  Interventions: Procedure: hernia repair

INTERVENTIONS:
Procedure: hernia repair — different methods for hernia repair

SUMMARY:
ventral hernias are defects of the anterior abdominal wall, which can be congenital or acquired including epigastric, umbilical and incisional hernia. Umbilical hernias represent a common surgical problem in cirrhotic patient with ascites with 20% incidence. This work was deigned to assess outcome of different techniques of closure of ventral hernias in cirrhotic patients.

DETAILED DESCRIPTION:
Ventral hernias are defects of the anterior abdominal wall, which can be congenital or acquired including epigastric, umbilical and incisional hernia. Incisional ventral hernia is a frequent complication of laparotomy that occurs in up to 11 % of surgical abdominal wounds

Umbilical hernia represent a common surgical problem in cirrhotic patient with ascites with 20% incidence.Factors that play role in occurance of umbilical hernia in cirrhotic patient with ascites patients is chronic increased intra-abdominal pressure, recanalization of the left umbilical vein, muscle wasting and fascial weakening from nutritional deficiencies (3,4).

Most of interventions for umbilical herniorrhaphy in cirrhotic patients with ascites done in emergency setting due to the concept of high perioperative morbidity and mortality rates in those patients. However, this strategy leads to a high risk of life-threatening complications such as incarceration and skin rupture.

ELIGIBILITY:
Inclusion Criteria:

* all cirrhotic patients with ventral hernia

Exclusion Criteria:

* hepatic encephalopathy

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: all patients with liver cirrhosis present with ventral hernias
Sampling Method: Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
ventral hernia repair | Baseline
  different technique for repair of ventral hernia